CLINICAL TRIAL: NCT00702611
Title: An Open Randomized Multicenter Clinical Investigation to Compare the Efficacy and Safety of Prednisone Plus Adacolumn® GMA Apheresis vs Prednisone Alone in the Treatment of Patients With Mild or Moderately Active Steroid Dependent Ulcerative Colitis
Brief Title: Efficacy Study of Granulocytapheresis Plus Steroids vs Steroids Alone in Active Steroid Dependant Ulcerative Colitis
Acronym: ATICCA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ada-UC-07-102
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Inflammatory Bowel disease; Steroid dependent; Adacolumn; Apheresis; Granulocyte Monocyte apheresis; GMA apheresis; Granulocytapheresis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Seven apheresis treatments over seven consecutive weeks (1/week) in conjunction with a starting dose of 40mg of oral prednisone per day at Week 00 for two weeks which will be tapered down to zero 5 mg/week within nine weeks
  Interventions: Device: Granulocyte Monocyte Apheresis (GMA-Apheresis)
- 2 (Active Comparator): Treatment with starting dose of 40mg of oral prednisone per day at Week 00 for two weeks and tapered down to zero 5 mg/week within nine weeks
  Interventions: Device: Granulocyte Monocyte Apheresis (GMA-Apheresis)

INTERVENTIONS:
Device: Granulocyte Monocyte Apheresis (GMA-Apheresis) — GMA Apheresis will be performed in a once per week during seven weeks only in experimental arm. Each apheresis will last 60 minutes at a blood flow rate of 30 ml/min.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the addition of GMA apheresis to steroid conventional treatment for achieving and maintaining remission in Active steroid dependant Ulcerative Colitis patients

DETAILED DESCRIPTION:
This is a multicenter randomized controlled trial which will compare the efficacy and safety of Adacolumn GMA apheresis plus oral steroids vs steroids alone in a strictly selected population of moderate to severe active steroid dependant Ulcerative Colitis patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years old
* Active ulcerative colitis with documented clinical symptoms and endoscopic findings
* Active disease defined as DAI (Mayo score) ≥ 4 and ≤10 with at least 1 point in flexible sigmoidoscopy
* Steroid dependency as defined by:

A. Inability to withdraw corticosteroids within three months of starting treatment, without recurrent active disease

B. appearance of relapse within 3 months after withdrawal of corticosteroids

* Colonic involvement with ulcerative colitis beyond 15cm of the anal verge
* Stable doses:A. Aminosalicylates for the last 4 weeks B. Prednisolone or equivalent dose ≤ 20 mg/day for the last 2 weeks C. Azathioprine or 6-mercaptopurine at stable dose for the last 12 weeks
* Signed informed consent form
* Agree to participate in the required follow-up visits
* Able to complete the diary

Exclusion Criteria:

* Febrile (> 38ºC)
* Evidence of toxic megacolon
* Anticipated need for surgery within 24 weeks
* Known obstructive diseases of the gastrointestinal system
* Proctocolectomy, total colectomy, ileostomy, stoma or ileal pouch-anal anastomosis
* A history of allergic reaction to heparin or heparin-induced thrombocytopenia
* A history of hypersensitivity reaction associated with an apheresis procedure or intolerance of apheresis procedures
* Requires a central venous access catheter for the apheresis treatments
* Known infection with enteric pathogens, pathogenic ova or parasites, C. difficile toxin or CMV
* Hypotension (systolic blood pressure <80 mmHg and/or diastolic blood pressure <50 mmHg) at screening visit only
* Uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >120 mmHg) despite medical therapy
* A history of myocardial infarction or unstable angina within the past 6 months
* A history of coronary artery bypass grafting surgery or angioplasty within the past 6 months
* Prosthetic heart valve, pacemaker or other permanent implant
* Severe cardiovascular or peripheral vascular disease, severe renal disease
* Liver disease defined as levels of SGOT [AST], SGPT [ALT] or alkaline phosphatase >2.5x the upper limit of the normal range for the laboratory performing test
* History of cirrhosis
* Known bleeding disorder (PT or PTT>1.5x the upper limit of the normal range for the laboratory performing the test), or concomitant anticoagulant therapy for purposes other than apheresis treatment
* Prior history suggestive of a hypercoagulable disorder, including 1 or more episodes of pulmonary embolism or deep vein thrombosis
* Known infection with Hepatitis B or C, or HIV
* Abnormal hematology parameters defined as severe anemia with hemoglobin <8.5g/dL, white blood cell count of <3,500/μl and a granulocyte count < 2,000/μl
* Fibrinogen level >700mg/dL
* Major surgery within the past 6 months
* Infection:Active infections less than 4 weeks from successful completion of antibiotic treatment for routine bacterial infectionFebrile viral infection within 4 weeks of entry into the clinical investigationLess than 12 weeks from conclusion of therapy for systemic fungal infections
* Malignancy within the past 2 years other than surgically cured skin carcinoma or cervical dysplasia (CIN I-II)
* History of dysplasia or carcinoma of the colon or lack of a complete colonoscopy in the last 12 months in patients with longstanding UC (> 10 años)
* Current drug or alcohol abuse
* Pregnant, lactating or planning to become pregnant during the course of the clinical investigation
* Used within the last 30 days an investigational drug, biologic or device or 5 half-lifes, if known, for any investigational drug or biologic
* Received cyclosporine or tacrolimus within the last 8 weeks
* Received infliximab within the last 8 weeks
* Fulminant ulcerative colitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in steroid free clinical remission defined by Mayo Score less or equal to 2 with no individual subscore >1 at week 24 | week 24

SECONDARY OUTCOMES:
Steroid free remission (assessed by Mayo score) | Week 12
Response at week 12 and 24 (defined by a decrease in Mayo Score > or = to 3 points | week 12 and week 24
Acute Phase reactants change at all lab analysis | 24 weeks
Rescue therapy requirements (new courses of steroids, cyclosporine, infliximab, or surgery) during study period | 24 weeks
Time to relapse | 24 weeks
· Clinical response according to the activity indexes Truelove & Witts, Powell Tuc, Rachmiliewitz (Clinical Activity Index), Lichtiger (Modified Truelove & Witts Severity Index), Walmsley (Simple Clinical Colitis Index | 24 weeks
Clinical remission and response at weeks 12 and 24 analysed according to concomitant use of immunosupressants | 24 weeks
Adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julian Panes, Ph D, Principal Investigator — Hospital Clinic i Provincial Barcelona; Joaquín Hinojosa, Ph D, Study Chair — Geteccu President; Daniel Ginard, MD, Study Director — Hospital Son Dureta Palma de Mallorca; Eugeni Domenech, Ph D, Principal Investigator — Germans Trias i Pujol Hospital; Raul Lafuente, MD, Principal Investigator — Otsuka Pharmaceutical S.A.; Fernando Magro, PhD, Principal Investigator — Hospital San Joao, Oporto; Vito Annesse, Ph D, Principal Investigator — Casa Sollievo de la Sofferenza, Italy
Locations (48):
- Medical University of Vienna, Vienna, Austria
- Germany (2):
  - Katolische Kliniken Ruhrhalbinsel, Essen
  - Markus-Krankenhaus, Frankfurt
- Italy (9):
  - Policlinico di Bari, Bari
  - Ospedale di Belluno, Belluno
  - Azienda Ospedaliero-Universitaria di Careggi, Florence
  - L'Azienda Unità Sanitaria Locale di Forlì, Forlì
  - Istituto Policlinico S. Donato, Milan
  - Policlinico di Padova, Padua
  - Policlinico Universitario Tor Vergata, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Casa Sollievo della Sofferenza, Istituto di Ricovero e Cura a Carattere Scientifico, Opera di San Pio da Pietrelcina, San Giovanni Rotondo
- Portugal (7):
  - Hospital da Universidade de Coimbra, Coimbra
  - Hospital Santa Maria, Lisbon
  - Instituto Portuges Oncologia Lisboa Francisco Gentil, Lisbon
  - Hospital Geral Santo Antonio, Porto
  - Hospital de Sao Joao, Porto
  - Hospital de Sao Bernardo, Setúbal
  - Hospital Sao Teotonio, Viseu
- Spain (29):
  - Complejo Hspitalario Universitario Santiago de Compostela, Santiago de Compostela, A Coruña
  - Complejo Universitario de Albacete, Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital General de Elche, Elche, Alicante
  - Complejo Hospitalario Reina Sofía, Córdoba, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital de Galdakano, Galdakao, Bilbao
  - Hospital Son Dureta, Palma de Mallorca, Comunidad Balear
  - Complejo Hospitalario Universitario Juan Canalejo, A Coruña, Galicia
  - Hospital Josep Trueta, Girona, Girona
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Leon, León, Leon
  - Clínica Puerta de Hierro, Madrid, Madrid
  - Hospital Fundación de Alcorcón, Madrid, Madrid
  - Hospital Universitario Clínico de San Carlos, Madrid, Madrid
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Puerto de Sagunto, Sagunto, Valencia
  - Hospital de Manises, Valencia, Valencia
  - Hospital Insular de Las Palmas, Las Palmas de Gran Canaria
  - Hospital Costa del Sol, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital do Meixoeiro, Vigo

REFERENCES:
- See also: Official web page of the GETECCU group — http://www.geteccu.org/